CLINICAL TRIAL: NCT00321789
Title: A Patient-Spouse Intervention for Self-Managing High Cholesterol
Acronym: CouPLES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: IIR 05-273
Record Dates: First submitted 2006-05-03; First posted 2006-05-04 (Estimated); Results first posted 2014-09-26 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2014-08

CONDITIONS: Hypercholesterolemia
Keywords: self care; social support
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spouse-assisted intervention (Experimental): Couples assigned to this arm received nine monthly phone calls from a nurse. The patient created goals and action plans related to diet, exercise, patient-provider communication, or medication adherence. The spouse developed a plan to support patient goal achievement.
  Interventions: Behavioral: spouse-assisted intervention
- Usual care (No Intervention): Couples assigned to this arm received educational materials at baseline and usual care thereafter, with no contact from the study interventionist.

INTERVENTIONS:
Behavioral: spouse-assisted intervention — Couples assigned to this arm received nine monthly phone calls from a nurse. The patient created monthly goals and action plans related to diet, exercise, patient-provider communication, or medication adherence. The spouse created plans to support patient goal achievement.
  Arms: Spouse-assisted intervention

SUMMARY:
We examined the effect of a patient-spouse intervention to lower LDL-C by increasing patient treatment adherence. A randomized controlled trial compared a one-year, telephone-based patient-spouse intervention to usual care. The primary outcome was LDL-C measured three times (baseline, 6 months, 11 months); secondary outcomes were adherence to medication, diet, and exercise, also assessed at baseline, 6 months, and 11 months.

DETAILED DESCRIPTION:
Background: Background/Rationale: Coronary heart disease (CHD) is the leading cause of death in the United States, resulting in more than 500,000 heart attacks and another 500,00 deaths per year. More than 80% of veterans have > 2 risk factors for CHD, underscoring the need for intervention. One major modifiable risk factor for CHD is elevated low-density lipoprotein cholesterol (LDL-C). Despite the proven success of diet, exercise, and medication, LDL-C frequently is not at the optimum level, due in part to patient nonadherence. Therefore, interventions are needed to increase adherence, thereby lowering LDL-C.

Objectives: Objectives: We examined the effect of a patient-spouse intervention to lower LDL-C by increasing patient treatment adherence. The primary hypothesis was that patients enrolled in a telephone-based, spouse-assisted intervention will experience a clinically meaningful 7% reduction in LDL-C. The secondary hypotheses were that patients who receive the intervention would show a significant increase in adherence to medication, diet, and exercise.

Methods: In a 3-year study, a randomized controlled trial compared a 10-month, telephone-based, spouse-assisted intervention to usual care. Married patients with above-goal LDL-C and their spouses were consented, completed a baseline assessment, and then were randomly assigned to the intervention or usual care arm. Month 1 involved an educational call delivered to patients and spouses. Months 2-10 (except month 6) involved monthly goal setting calls delivered to patients and calls focused on increasing social support to spouses. The patient phone call will always preceded the spouse phone call. At 6 and 11 months, LDL-C and adherence were re-assessed. The primary outcome was LDL-C measured three times (baseline, 6 months, 11 months); secondary outcomes were adherence to medication, diet, and exercise, also assessed at baseline, 6 months, and 11 months. Descriptive statistics were computed for all study variables within each study arm. Mixed effects models were used to evaluate the intervention's effect on the primary and secondary outcomes at 11 months. We also calculated intervention cost.

Status: Enrollment began in Fall, 2007 and was completed in July of 2009.

Impact: Elevated LDL-C is a major risk factor for CHD, stroke, and peripheral vascular disease, all of which are common among veterans. The expected increase in prevalence of CHD over the next several decades will result in an increased burden for both veterans and the VA health care system. Despite the known risk of hypercholesterolemia, many veterans have suboptimal LDL-C levels. As the latest evidence and recommendations suggest that these goals should be even lower, interventions to assist patients to lower LDL-C increasingly will be needed. The VA considers the reduction of LDL-C an important goal, as indicated by the major effort of the Ischemic Heart Disease Quality Enhancement Research Initiatives (QUERI). This study is important because (1) it addresses a highly prevalent risk factor for CHD among veterans; (2) it proposes a potentially low-cost method for improving LDL-C levels, which in turn could reduce VA healthcare costs; (3) the intervention is practical and could be disseminated easily in the VA healthcare system if proven effective; and (4) this intervention provides a model for self-management of other chronic diseases, such as diabetes and hypertension.

ELIGIBILITY:
Inclusion Criteria:

* veteran
* elevated baseline low-density lipoprotein cholesterol level
* married

Exclusion Criteria:

* no telephone number;
* spouse unwilling to participate;
* patient or spouse cognitively impaired, unable to communicate via telephone, living in nursing home or receiving home health care, or refuses to provide informed consent;
* hospitalized past 3 months;
* survival prognosis less than 1 year;
* active psychosis or dementia; no primary care physician at VA;
* no medical visit to VA in past year;
* enrolled in another study focusing on lifestyle changes

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2007-09; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corrine I. Voils, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

REFERENCES:
- [Result] Voils CI, Yancy WS Jr, Weinberger M, Bolton J, Coffman CJ, Jeffreys A, Oddone EZ, Bosworth HB. The trials and tribulations of enrolling couples in a randomized, controlled trial: a self-management program for hyperlipidemia as a model. Patient Educ Couns. 2011 Jul;84(1):33-40. doi: 10.1016/j.pec.2010.06.005. Epub 2010 Jul 5. PMID 20599337
- [Result] Voils CI, Yancy WS Jr, Kovac S, Coffman CJ, Weinberger M, Oddone EZ, Jeffreys A, Datta S, Bosworth HB. Study protocol: Couples Partnering for Lipid Enhancing Strategies (CouPLES) - a randomized, controlled trial. Trials. 2009 Feb 6;10:10. doi: 10.1186/1745-6215-10-10. PMID 19200384
- [Result] Voils CI, Coffman CJ, Yancy WS Jr, Weinberger M, Jeffreys AS, Datta S, Kovac S, McKenzie J, Smith R, Bosworth HB. A randomized controlled trial to evaluate the effectiveness of CouPLES: a spouse-assisted lifestyle change intervention to improve low-density lipoprotein cholesterol. Prev Med. 2013 Jan;56(1):46-52. doi: 10.1016/j.ypmed.2012.11.001. Epub 2012 Nov 9. PMID 23146744
- [Result] Gallagher P, Yancy WS Jr, Jeffreys AS, Coffman CJ, Weinberger M, Bosworth HB, Voils CI. Patient self-efficacy and spouse perception of spousal support are associated with lower patient weight: baseline results from a spousal support behavioral intervention. Psychol Health Med. 2013;18(2):175-81. doi: 10.1080/13548506.2012.715176. Epub 2012 Sep 10. PMID 22963235
- [Result] King HA, Jeffreys AS, McVay MA, Coffman CJ, Voils CI. Spouse health behavior outcomes from a randomized controlled trial of a spouse-assisted lifestyle change intervention to improve patient low-density lipoprotein cholesterol. J Behav Med. 2014 Dec;37(6):1102-7. doi: 10.1007/s10865-014-9559-4. Epub 2014 Mar 2. PMID 24584818
- [Result] Sperber NR, Sandelowski M, Voils CI. Spousal support in a behavior change intervention for cholesterol management. Patient Educ Couns. 2013 Jul;92(1):121-6. doi: 10.1016/j.pec.2013.02.015. Epub 2013 Mar 27. PMID 23541217

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Couples enrolled in the intervention arm received educational materials at baseline, followed by eight monthly phone calls from a study nurse. Each month, the patient participant created goals and action plans related to diet, exercise, patient-provider communication, or medication adherence. Following the patient call, the spouse participant was informed of the patient's goals and action plans developed a support plan to help the patient achieve his or her goal.
- Usual Care: Couples assigned to usual care received educational materials at baseline and usual care to the patient thereafter, with no contact from the study interventionist.
Period: Overall Study
Arm/Group | Intervention | Usual Care
Started | 127 | 128
Completed | 112 | 112
Not Completed | 15 | 16
Not completed — Lost to Follow-up | 4 | 7
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Protocol Violation | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Usual Care | Total
Number analyzed (Participants) | 127 | 128 | 255
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (12.3) | 61.0 (12.2) | 61.3 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 13
  Male | 117 | 125 | 242
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 35 | 43 | 78
  White | 82 | 81 | 163
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 3 | 12
Region of Enrollment [Number; unit: participants]
  United States | 127 | 128 | 255
Education [Number; unit: participants]
  8th grade or less | 2 | 2 | 4
  some high school | 4 | 6 | 10
  high school degree or equivalent | 26 | 20 | 46
  some college or vocational training, no degree | 34 | 35 | 69
  Associate's degree | 23 | 21 | 44
  Bachelor's degree | 19 | 28 | 47
  Graduate or professional degree | 16 | 15 | 31
  not reported | 3 | 1 | 4
Employment status [Number; unit: participants]
  working full time | 46 | 58 | 104
  working part time | 19 | 10 | 29
  unemployed, searching for work | 5 | 5 | 10
  unemployed, not searching for work | 3 | 2 | 5
  retired | 43 | 47 | 90
  disabled | 8 | 5 | 13
  not reported | 3 | 1 | 4
High risk for cardiovascular event based on Framingham score [Number; unit: participants]
  high risk | 25 | 19 | 44
  low or moderate risk | 102 | 109 | 211
number of participants who met goal for low-density lipoprotein cholesterol at baseline [Number; unit: participants] — Goal is determined by 2003 National Cholesterol Education Program guidelines. Goal could be 160mg/dL for low risk (no coronary heart disease (CHD), 0-1 risk factor); 130 mg/dL for medium risk (no CHD, at least 2 risk factors); or 100 mg/dL for high risk (CHD and risk equivalents including diabetes, atherosclerotic disease, and multiple risk factors that confer a 10-year risk for CHD >20% per Framingham score).
  participants
    met goal | 45 | 62 | 107
    did not meet goal | 82 | 66 | 148
number of participants prescribed cholesterol medication at baseline [Number; unit: participants]
  taking cholesterol medication | 62 | 57 | 119
  not taking cholesterol medication | 65 | 71 | 136
Missed at least one dose of cholesterol medication in previous 30 days at baseline [Number; unit: participants] — Based on self-report to a single item querying whether participants missed doses in the previous 30 days.
  participants
    missed at least one dose | 31 | 28 | 59
    did not miss at least one dose | 31 | 29 | 60
    not relevant (not taking medication) | 65 | 71 | 136

OUTCOME MEASURES:

1. Primary Outcome: Low-density Lipoprotein Cholesterol
Description: assessed with non-fasting blood test
Time Frame: 11-month follow-up
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 127 | 128
mg/dL | 123.6 (25.6) | 115.3 (27.8)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority or Other; p = 0.44, Mixed Models Analysis; Model was adjusted for a priori race and cardiovascular disease risk level strata; Mean Difference (Final Values) = 2.3, 95% CI 2-sided [-3.6 to 8.3]

2. Secondary Outcome: Caloric Intake
Description: Self-reported, assessed via Block Brief Food Frequency Questionnaire (FFQ).
Time Frame: 11-month follow-up
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 115 | 109
kcal/day | 1175.3 (578.8) | 1253.9 (575.0)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority or Other; p = 0.03, Mixed Models Analysis; Based on log-transformed values. Model was adjusted for a priori race and cardiovascular disease risk level strata; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-0.23 to -0.01]

3. Secondary Outcome: Saturated Fat (Grams/Day)
Description: Self-reported, assessed via Block Brief Food Frequency Questionnaire (FFQ).
Time Frame: 11-month follow-up
Measure: Mean (Standard Deviation); unit: grams per day
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 115 | 109
grams per day | 15.1 (8.9) | 17.4 (9.8)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority or Other; p = 0.02, Mixed Models Analysis; Based on log-transformed values. Model was adjusted for a priori race and cardiovascular disease risk level strata; Mean Difference (Net) = -0.16, 95% CI 2-sided [-0.29 to -0.02]

4. Secondary Outcome: Total Fat (Grams/Day)
Description: Self-reported, assessed via Block Brief Food Frequency Questionnaire (FFQ).
Time Frame: 11-month follow-up
Measure: Mean (Standard Deviation); unit: grams per day
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 115 | 109
grams per day | 46.5 (25.6) | 54.2 (31.1)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority or Other; p = 0.02, Mixed Models Analysis; Based on log-transformed values. Model was adjusted for a priori race and cardiovascular disease risk level strata; Mean Difference (Net) = -0.16, 95% CI 2-sided [-0.29 to -0.03]

5. Secondary Outcome: Cholesterol Intake
Description: Self-reported, assessed via Block Brief Food Frequency Questionnaire (FFQ).
Time Frame: 11-month follow-up
Measure: Mean (Standard Deviation); unit: milligrams per day
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 115 | 109
milligrams per day | 152.1 (97.4) | 175.5 (117.1)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority or Other; p = 0.11, Mixed Models Analysis; Based on log-transformed values. Model was adjusted for a priori race and cardiovascular disease risk level strata; Mean Difference (Net) = -0.13, 95% CI 2-sided [-0.30 to 0.03]

6. Secondary Outcome: Fiber Intake
Description: Self-reported, assessed via Block Brief Food Frequency Questionnaire.
Time Frame: 11-month follow-up
Measure: Mean (Standard Deviation); unit: grams per day
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 115 | 109
grams per day | 13.2 (6.3) | 11.9 (5.7)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority or Other; p = 0.26, Mixed Models Analysis; Based on log-transformed values. Model was adjusted for a priori race and cardiovascular disease risk level strata; Mean Difference (Net) = 0.07, 95% CI 2-sided [-0.06 to 0.20]

7. Secondary Outcome: Frequency of Moderate Intensity Physical Activity
Description: Self-reported via Community Health Activities Model Program for Seniors questionnaire.
Time Frame: 11-month follow-up
Measure: Median (Inter-Quartile Range); unit: times per week
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 127 | 128
times per week | 10 [6 to 14] | 10 [4 to 16]
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority or Other; p = 0.06, generalized estimating equations; Based on log-transformed values. Model was adjusted for a priori race and cardiovascular disease risk level strata; incident rate ratio = 1.2, 95% CI 2-sided [1.0 to 1.5]

8. Secondary Outcome: Duration of Moderate Intensity Physical Activity
Description: Self-reported via Community Health Activities Model Program for Seniors questionnaire.
Time Frame: 11-month follow-up
Measure: Median (Inter-Quartile Range); unit: hours per week
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 127 | 128
hours per week | 7.3 [3.9 to 10.8] | 7.8 [3.5 to 12.3]
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority or Other; p = 0.37, generalized estimating equations; Model adjusted for a priori race and cardiovascular disease risk category; incident rate ratio = 1.1, 95% CI 2-sided [0.9 to 1.4]

9. Secondary Outcome: Total Fat (%)
Description: Self-reported, assessed via Block Brief Food Frequency Questionnaire (FFQ).
Time Frame: 11-month follow-up
Measure: Mean (Standard Deviation); unit: percentage of calories
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 115 | 109
percentage of calories | 35.4 (7.3) | 38.2 (9.1)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority or Other; p = 0.04, Mixed Models Analysis; Model adjusted for a priori race and cardiovascular disease risk category; Mean Difference (Net) = -2.11, 95% CI 2-sided [-4.13 to -0.09]

10. Secondary Outcome: Saturated Fat (%)
Description: Self-reported, assessed via Block Brief Food Frequency Questionnaire (FFQ).
Time Frame: 11-month follow-up
Measure: Mean (Standard Deviation); unit: percentage of calories
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 115 | 109
percentage of calories | 11.4 (2.8) | 12.3 (2.9)
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority or Other; p = 0.09, Mixed Models Analysis; Model adjusted for a priori race and cardiovascular disease risk category; Mean Difference (Net) = -0.64, 95% CI 2-sided [-1.38 to 0.10]

11. Secondary Outcome: Number of Participants With Goal LDL-C
Description: Assessed via non-fasting blood test. Goal is determined by 2003 National Cholesterol Education Program guidelines. Goal could be 160mg/dL for low risk (no coronary heart disease (CHD), 0-1 risk factor); 130 mg/dL for medium risk (no CHD, at least 2 risk factors); or 100 mg/dL for high risk (CHD and risk equivalents including diabetes, atherosclerotic disease, and multiple risk factors that confer a 10-year risk for CHD >20% per Framingham score).
Time Frame: 11-month follow-up
Measure: Number; unit: participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 127 | 128
participants | 57 | 62
Statistical Analysis 1: Comparison: Intervention vs Usual Care; Test type: Superiority or Other; p = 0.87, Regression, Logistic; Model adjusted for a priori race and cardiovascular disease risk category; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.6 to 1.7]

12. Secondary Outcome: Number of Participants Prescribed Cholesterol Medication
Description: This was assessed via electronic medical record abstraction. Results could not be modeled statistically due to missing data/small cell sizes (i.e., not all participants had a prescription for medication because this was not an inclusion criterion).
Time Frame: 11-month follow-up
Measure: Number; unit: participants
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 127 | 128
participants | 56 | 56

ADVERSE EVENTS:
Time Frame: 11 months
Arm/Group | Intervention | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/127 | 1/128
Other Adverse Events (participants affected / at risk) | 0/127 | 0/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=127) | Usual Care (N=128)
death (General disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The dietary measure underestimates dietary intake but should not invalidate differences between groups or across time. Sample size for dietary analyses was reduced due to missing data, but non-responders did not differ on measured characteristics.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes